CLINICAL TRIAL: NCT03110094
Title: Investigation of Immunological and Pharmacological Factors for Response to Adalimumab in Rheumatoid Arthritis, With Analysis of CD4 + Follicular Helper T Subpopulations
Brief Title: Investigation of Immunological and Pharmacological Factors for Response to Adalimumab in Rheumatoid Arthritis
Acronym: PROMETHEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC17_3063_PROMETHEE
Record Dates: First submitted 2017-03-10; First posted 2017-04-12 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rheumatoid arthritis - Adalimumab (Other)
  Interventions: Other: Adalimumab
- Healthy volunteer (Other)
  Interventions: Other: Healthy volunteers

INTERVENTIONS:
Other: Adalimumab — It will be an interventional study with minimal risks and constraints, prospective, mono-centric, in current care. Patient management will not be changed during the study. It will be taken at two different tracking points (M0 and M3) 4 additional tubes and use of surplus articular fluid (M0 and M3).
  Other Names: Additional Biological Sample
  Arms: Rheumatoid arthritis - Adalimumab
Other: Healthy volunteers — Collection of 2 tubes of blood. The values of the quantitative study of lymphocyte subpopulations will be compared to those obtained from healthy blood donors to define the standards used in this study.
  Other Names: Recovery of blood tubes during a donation
  Arms: Healthy volunteer

SUMMARY:
Interventional study with minimal risks and constraints, prospective, mono-centric.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory disease with synovial tropism, characterized by joint pain and swelling, secondary to inflammation of the synovial membrane and which can lead to joint destruction, with the risk of a major functional disability. Biological treatments have revolutionized its management over the past 15 years. However, they are not effective in all patients, they are expensive, and are not without side effects sometimes severe.

Currently, there is no predictive factor for response to biotherapy beyond the severity criteria of rheumatoid arthritis (presence of erosions, presence of anti-Citrullinated Protein Antibody (ACPA), importance of biological and clinical inflammation ).

The role of T lymphocytes and B lymphocytes has been widely studied in rheumatoid arthritis. The activity of rheumatoid arthritis is associated with a Th1 and Th17 type CD4 + T polarization, with pro-inflammatory cytokine production and decreased Treg activity.

In recent years, a population of CD4 + T lymphocytes, Tfh (T follicular helper cells) has been demonstrated and seems likely to play an important role in the pathogenesis of rheumatoid arthritis. Physiologically these cells were initially described in the secondary lymphoid organs where they are essential for the survival and differentiation of B lymphocytes into antibody-secreting cells. More recently, they have been described in the blood (c Tfh for circulating T follicular helper cells) and appear to be a reflection of Tfh activity in tissues.

Several studies have focused on c Tfh in rheumatoid arthritis. A significantly higher level of c Tfh was observed in rheumatoid arthritis than in healthy controls. A significant positive correlation was also observed between the level of c Tfh and the titre of ACPA and between the rate of c Tfh and the activity of the rheumatoid arthritis, measured by the Disease Activity Score (DAS). However, each research group characterized the c Tfh t with different markers, which limits the comparison of the different results obtained.

The rate of c Tfh also appears to be influenced by treatments. In a Chinese rheumatoid arthritis study, the level of c Tfh was analyzed before and after one month of treatment with Methotrexate and phytotherapy with Tripterygium wilfordii. The rate of cTfh had significantly decreased in the responders whereas it had not decreased in the non responders. All of these first results, observed in a limited number of patients, are in favor of a relationship between the level of c Tfh and the activity and / or severity of rheumatoid arthritis, and on the other hand, suggest that variations in c Tfh might be related to response to treatment.

The analysis of peripheral blood lymphocyte cells has the advantage of ease of access, by simple venipuncture. However, these cells do not always accurately reflect the populations present within the synovial membrane. The analysis of the cells of the synovial membrane requires the realization of a biopsy, invasive gesture and incompatible with the practice in routine care. The analysis of the cells of the articular fluid would make it possible to better apprehend the resident populations of the synovial membrane without generating an over-risk for the patient. Indeed the gesture of joint puncture is justified in case of effusion by the diagnosis (to eliminate an infection) and therapeutic (to carry out if necessary an injection of corticosteroids). Rheumatoid arthritis joint fluids are inflammatory, defined by a number of nucleated elements greater than 2000 / mm3. The flow cytometry study, using the same phenotypic markers as those used for peripheral blood analysis, in patients in thrust will allow comparison of lymphocyte blood subpopulations and joint fluid.

The existence of a predictive serum biomarker of response or nonresponse to anti-TNFα therapy would improve the management of patients by avoiding delaying the use of potentially more effective treatment in patients Priori non-responders to an anti-TNF α biotherapy. If approximately 25% of the patients are not responding to a first biotherapy, it would be interesting to be able to identify them upstream, using a predictive marker, in order to orient them early to another therapy.

Remote infrared infrared spectroscopy, using a chalcogenide glass optical fiber, allows the study of the functional groups of the molecules present in a biological sample. It showed its ability, through the demonstration of changes in spectroscopic profiles, to discriminate samples representing physiological and pathological situations. This method has shown an interest in the early diagnosis of septic arthritis from joint puncture fluid, for the diagnosis of RA from serum and for staging of hepatic steatosis from serum.

The objective of this work is to investigate whether the quantitative and / or qualitative variations of different lymphocyte subpopulations (especially Tfh) in a rheumatoid arthritis population treated with the same anti-TNF alpha (Tumor Necrosis Factor ), Adalimumab, are likely to influence the response or non-response to treatment at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis diagnosed according to EULAR 2010 criteria (European League Against Rheumatism);
* Active rheumatoid arthritis, defined by DAS 28> 3.2;
* Corticotherapy systemic ≤ 15mg /day, stable for ≥ 15 days;
* Refractory or intolerant rheumatoid arthritis with at least one chemical background treatment;
* Previous biological treatment stopped for ≥ 3 months for monoclonal antibodies (except Rituximab) and 15 days for Etanercept;
* Patients who have given written informed consent.
* For healthy volunteers: subjects aged 18 coming to the French blood establishment of Rennes for a donation of blood

Exclusion Criteria:

* Patient minor;
* Presence of a contraindication to biological treatment;
* Previous treatment with Rituximab;
* Vaccination or surgery in the month preceding the study or planned within 3 months of inclusion;
* Patient not affiliated to social security;
* Major persons subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of their liberty.
* For healthy volunteers: Minor subject ; Subject not affiliated with social security ; Major persons subject to legal protection (legal safeguards, guardianship, tutorship), persons deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Patient responding or not responding to treatment with Adalimumab at 6 months defined by a value of Disease Activity Score 28 (DAS 28) ≤ 3.2. | 6 months
  Disease Activity Score 28 (DAS 28) calculated in every patients after clinical examination.

SECONDARY OUTCOMES:
Patient responding or not responding to treatment with Adalimumab at 1 year defined by a value of Disease Activity Score 28 (DAS 28) ≤ 3.2. | 12 months
  Disease Activity Score 28 (DAS 28) calculated in every patients after clinical examination.
Patient responding or not responding to treatment with Adalimumab at 6 months and 1 year defined by the SDAI scores | 6 and 12 months
  SDAI score will be calculated in every patients after clinical examination.
Patient responding or not responding to treatment with Adalimumab at 6 months and 1 year defined by the CDAI scores | 6 and 12 months
  CDAI score will be calculated in every patients after clinical examination.
Patient responding or not responding to treatment with Adalimumab at 6 months and 1 year defined by the HAQ scores | 6 and 12 months
  HAQ will be calculated in every patients after self-assessment questionnaire.
Residual plasmatic Adalimumab concentration | 3, 6 and 12 months
Count of Anti-Adalimumab antibody | 3, 6 and 12 months
Second derivative spectrometric profiles | Baseline and 3 monts
  Serum and joint fluid

CONTACTS AND LOCATIONS:
Overall Officials: Aleth Perdriger, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No